CLINICAL TRIAL: NCT01419964
Title: Phase III, Multicenter, Randomized, Double-blind, Placebo-controlled Parallel Group Study of the Efficacy and Safety of ACH24 in the Treatment of Vitiligo
Brief Title: Efficacy and Safety of ACH24 in the Treatment of Vitiligo
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The Brazilian regulatory agency - ANVISA has requested the cancellation of the phase 3 study for conducting a phase 1 study first.
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACH-VTL-03(09/11)
Record Dates: First submitted 2011-08-17; First posted 2011-08-19 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Vitiligo
Keywords: Vitiligo; Macular depigmentation; Stachytarpheta cayensensis
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 01 (Experimental): ACH24
  Interventions: Drug: Group 01
- Group 02 (Placebo Comparator): Placebo
  Interventions: Drug: Group 02

INTERVENTIONS:
Drug: Group 01 — ACH24
  Other Names: ACH24
  Arms: Group 01
Drug: Group 02 — Placebo
  Other Names: PLACEBO
  Arms: Group 02

SUMMARY:
This is a multicenter clinical trial, phase III, randomized, placebo-controlled, parallel group, enroll 94 patients, to assess the efficacy of ACH24 in the repigmentation of achromatic areas in patients with vitiligo.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of ACH24 compared to placebo in the treatment of vitiligo.The present study aims to register a new product in the country, the ACH24 for the treatment of vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged between 18 and 65 years, remaining the feasibility of a legal guardian in accordance with need, able to understand and provide written informed consent and able to allow compliance at the treatment and the requirements of the protocol;
* Presence of generalized vitiligo;
* Able to comprehend and willing to provide written informed consent in accordance with institutional and regulatory guidelines.

Exclusion Criteria:

* Patients with:

  * Inflammatory diseases;
  * Alopecia Areata;
  * Diabetes Type I;
  * Asthma;
  * Collagen disease;
  * Atopic dermatitis;
  * Psoriasis;
  * Autoimmune thyroid disease (self reported). ¬ Thyroid problems (represents 15% of people with vitiligo), exclude only those who need to do treatment with corticosteroid or immunosuppressive.
* Women of childbearing age who had tested positive for pregnancy, or who do not use acceptable contraceptive method, or do not agree to practice reliable contraception during the study;
* Woman in pregnancy or lactation period;
* Known allergic reaction against the phytomedicine as assessed by medical history;
* Patient that is taking any prohibited medication (Item 9.3);
* Participation in last one year of clinical protocols, unless it can be direct benefit to subject;
* Any finding of clinical observation (anamnesis and physical exam) laboratory abnormality (eg, blood glucose, blood count), disease (for example, liver, cardiovascular system, lung) or therapy that, in opinion of the investigator, may endanger the subject or interfere with the endpoints of study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Repigmentation of the affected area assessed by VASI (vitiligo area scoring index). | Baseline compared to the end of 18 months of treatment
  It is considered successful treatment a repigmentation of greater than or equal to 50% of the affected area assessed by VASI (vitiligo area scoring index).

SECONDARY OUTCOMES:
Quality of life questionnaire | Baseline and each 12 weeks of treatment (V0, V3, V6, V9, V12, V15, V18)
  Dermatology Life Quality Index (DLQI)
Safety descriptive about occurence of adverse events, evaluation of results of general physical examination. | Will be evaluated during whole study, at the baseline and after 18 months of treatment
  Collection of safety data throughout the whole study period

CONTACTS AND LOCATIONS:
Overall Officials: CAIO CASTRO, PHYSICIAN, Principal Investigator — PUNTIFÍCIA UNIVERSIDADE CATÓLICA
Locations (1):
- Irmandade da Santa Casa de Misericórdia de Curitiba, Curitiba, Paraná, Brazil